CLINICAL TRIAL: NCT00002851
Title: PHASE III RANDOMISED TRIAL INVESTIGATING THE ROLE OF INTERNAL MAMMARY AND MEDIAL SUPRACLAVICULAR (IM-MS) LYMPH NODE CHAIN IRRADIATION IN STAGE I-III BREAST CANCER
Brief Title: Lymph Node Radiation Therapy in Patients With Stage I, Stage II, or Stage III Breast Cancer That Has Been Surgically Removed
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065094; EORTC-10925; EORTC-22922
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2004-12

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Chemotherapy, Adjuvant

INTERVENTIONS:
Procedure: adjuvant therapy
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Radiation therapy may kill any tumor cells remaining after surgery.

PURPOSE: This randomized phase III trial is studying radiation therapy to see how well it works compared to no further therapy in treating women with stage I, stage II, or stage III breast cancer that has been surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of irradiation of the homolateral internal mammary and medial supraclavicular lymph node chains vs no further therapy on survival, disease-free survival, metastasis-free survival, and cause of death in women with resected stage I/II/III breast cancer.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by participating institution, tumor location, type of prior breast surgery, pathologic T and N stage, menopausal status, and time sequence of radiotherapy and adjuvant chemotherapy. Patients are randomized to 1 of 2 arms.

* Arm I: Patients receive no nodal irradiation.
* Arm II: Patients receive irradiation of the internal mammary and medial supraclavicular lymph node chains delivered at 1 fraction per day, 5 sessions per week, for a total of 25 fractions over 5 weeks. Radiotherapy must begin no later than 8 weeks after surgery. If adjuvant chemotherapy is given, radiotherapy begins within 6 weeks after the last course of chemotherapy and within 8 months after surgery.

Patients are followed at least yearly after randomization for up to 20 years.

PROJECTED ACCRUAL: A total of 4,000 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unilateral adenocarcinoma of the breast
* Stage I/II/III (Tx, T0-3, N0-2) disease in one of the following categories or multifocal tumors if one of the foci is in agreement with the following:

  * Centrally or medially located with any lymph node status

    * Central location defined as underlying the areola
    * Medial location defined as at least partial involvement of upper or lower medial quadrant of breast
  * Externally located with axillary node involvement
* Prior mastectomy or breast-conserving surgery and axillary dissection required

  * Sentinel node procedure as axillary intervention without further axillary surgery is allowed
  * No prior internal mammary chain dissection
  * No upper inner lesion treated with breast-conserving surgery that precludes sparing of internal mammary lymph node chain from radiotherapy volume

    * Decision at radiation oncologist's discretion
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 75 and under

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No prior cardiac disease

Other:

* No prior malignancy except adequately treated nonmelanomatous skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* Concurrent enrollment in other randomized trials allowed

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 1996-07

CONTACTS AND LOCATIONS:
Overall Officials: Walter F. Van den Bogaert, MD, PhD — University Hospital, Gasthuisberg; H. Struikmans, MD, PhD — Medisch Centrum Haaglanden Westeinde; Alain Fourquet, MD — Institut Curie; Harry Bartelink, MD, PhD — The Netherlands Cancer Institute
Locations (48):
- Belgium (6):
  - Ziekenhuis Network Antwerpen Middelheim, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - Hopital de Jolimont, Haine-Saint-Paul
  - Cazk Groeninghe - Campus Maria's Voorzienigheid, Kortrijk
  - U.Z. Gasthuisberg, Leuven
  - Algemeen Ziekenhuis Sint-Augustinus, Wilrijk
- Institute of Oncology - Clinical Center University of Sarajevo, Sarajevo, Bosnia and Herzegovina
- Chile (2):
  - Instituto de Radiomedicina, Santiago
  - Clinica Alemana, Santiago
- France (11):
  - CHR de Besancon - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Service Cancerologie Polyclinique Clairval, Marseille
  - Centre Antoine Lacassagne, Nice
  - Centre Eugene Marquis, Rennes
  - Centre Hospitalier Universitaire Henri Mondor, Strasbourg
  - Centre Leon Berard, Strasbourg
  - Centre Paul Strauss, Strasbourg
  - Institut Gustave Roussy, Strasbourg
- Germany (7):
  - Charite - Campus Charite Mitte, Berlin
  - Robert Roessle Comprehensive Cancer Center at University of Berlin - Charite Campus Buch, Berlin
  - Klinik I fuer Innere Medizin, Cologne
  - University of Erlangen-Nuremberg, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Goettingen, Göttingen
  - Universitaetsklinikum Tuebingen, Tübingen
- Israel (2):
  - Rambam Medical Center, Haifa
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (2):
  - Ospedale Sant Anna, Como
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa (Genova)
- Netherlands (9):
  - Medisch Centrum Haaglanden, 's-Gravenhage (Den Haag, the Hague)
  - Academisch Medisch Centrum, Amsterdam
  - Streekziekenhuis Gooi-Noord, Blaricum
  - Radiotherapeutisch Instituut-(Riso), Deventer
  - Medisch Spectrum Twente, Enschede
  - Academisch Ziekenhuis Groningen, Groningen
  - Radiotherapeutisch Instituut Limburg-Maastricht, Maastricht
  - Dr. Bernard Verbeeten Instituut, Tilburg
  - Academisch Ziekenhuis Utrecht, Utrecht
- Medical University of Gdansk, Gdansk, Poland
- Instituto Portugues de Oncologia Centro do Porto, SA, Porto, Portugal
- Institut Catala D'Oncologia, Barcelona, Spain
- Switzerland (3):
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - UniversitaetsSpital, Zurich
- Istanbul University-Institute of Oncology, Istanbul, Turkey (Türkiye)
- Nottingham City Hospital NHS Trust, Nottingham, England, United Kingdom

REFERENCES:
- [Result] Matzinger O, Heimsoth I, Poortmans P, Collette L, Struikmans H, Van Den Bogaert W, Fourquet A, Bartelink H, Ataman F, Gulyban A, Pierart M, Van Tienhoven G; EORTC Radiation Oncology & Breast Cancer Groups. Toxicity at three years with and without irradiation of the internal mammary and medial supraclavicular lymph node chain in stage I to III breast cancer (EORTC trial 22922/10925). Acta Oncol. 2010;49(1):24-34. doi: 10.3109/02841860903352959. PMID 20100142
- [Result] Musat E, Poortmans P, Van den Bogaert W, Struikmans H, Fourquet A, Bartelink H, Kirkove C, Budach V, Pierart M, Collette L. Quality assurance in breast cancer: EORTC experiences in the phase III trial on irradiation of the internal mammary nodes. Eur J Cancer. 2007 Mar;43(4):718-24. doi: 10.1016/j.ejca.2006.11.015. Epub 2007 Jan 19. PMID 17240136
- [Result] Poortmans P, Kouloulias V, van Tienhoven G, Collette L, Struikmans H, Venselaar JL, Van den Bogaert W, Davis JB, Lambin P; EORTC Radiation Oncology and Breast Cancer Groups. Quality assurance in the EORTC randomized trial 22922/10925 investigating the role of irradiation of the internal mammary and medial supraclavicular lymph node chain works. Strahlenther Onkol. 2006 Oct;182(10):576-82. doi: 10.1007/s00066-006-1629-2. PMID 17013570
- [Result] Poortmans P, Kouloulias VE, Venselaar JL, Struikmans H, Davis JB, Huyskens D, van Tienhoven G, Hurkmans C, Mijnheer B, Van den Bogaert W. Quality assurance of EORTC trial 22922/10925 investigating the role of internal mammary--medial supraclavicular irradiation in stage I-III breast cancer: the individual case review. Eur J Cancer. 2003 Sep;39(14):2035-42. doi: 10.1016/s0959-8049(03)00455-6. PMID 12957458
- [Result] Poortmans PM, Venselaar JL, Struikmans H, Hurkmans CW, Davis JB, Huyskens D, van Tienhoven G, Vlaun V, Lagendijk JJ, Mijnheer BJ, De Winter KA, Van der Hulst MH, Van den Bogaert WF. The potential impact of treatment variations on the results of radiotherapy of the internal mammary lymph node chain: a quality-assurance report on the dummy run of EORTC Phase III randomized trial 22922/10925 in Stage I--III breast cancer(1). Int J Radiat Oncol Biol Phys. 2001 Apr 1;49(5):1399-408. doi: 10.1016/s0360-3016(00)01549-2. PMID 11286848
- [Result] Poortmans P, Van Den Bogaert W, Venselaar J, et al.: Quality assurance in EORTC trial 22922/10925 concerning internal mammary chain (IMC) irradiation: the dummy run. Radiother Oncol 48(suppl 1): A735, s186, 1998.
- [Result] Poortmans P, Van Den Bogaert W, Venselaar J, et al.: EORTC randomized phase III trials 22922/10925 investigating the role of internal mammary chain (IMC) irradiation in stage I-II breast cancer: a quality assurance report on the dummy run. Eur J Cancer 34(suppl 5): A257, s58, 1998.
- [Derived] Kaidar-Person O, Fortpied C, Hol S, Weltens C, Kirkove C, Budach V, Peignaux-Casasnovas K, van der Leij F, Vonk E, Valli M, Weidner N, Guckenberger M, Koiter E, Fourquet A, Bartelink H, Struikmans H, Poortmans P; EORTC Radiation Oncology and Breast Cancer Groups. The association of internal mammary and medial supraclavicular lymph node radiation technique with clinical outcomes: Results from the EORTC 22922/10925 randomised trial. Radiother Oncol. 2022 Jul;172:99-110. doi: 10.1016/j.radonc.2022.05.006. Epub 2022 May 12. PMID 35568284
- [Derived] Poortmans PM, Struikmans H, De Brouwer P, Weltens C, Fortpied C, Kirkove C, Budach V, Peignaux-Casasnovas K, van der Leij F, Vonk E, Valli M, vanTienhoven G, Weidner N, Noel G, Guckenberger M, Koiter E, vanLimbergen E, Engelen A, Fourquet A, Bartelink H; EORTC Radiation Oncology and Breast Cancer Groups. Side Effects 15 Years After Lymph Node Irradiation in Breast Cancer: Randomized EORTC Trial 22922/10925. J Natl Cancer Inst. 2021 Oct 1;113(10):1360-1368. doi: 10.1093/jnci/djab113. PMID 34320651
- [Derived] Poortmans PM, Weltens C, Fortpied C, Kirkove C, Peignaux-Casasnovas K, Budach V, van der Leij F, Vonk E, Weidner N, Rivera S, van Tienhoven G, Fourquet A, Noel G, Valli M, Guckenberger M, Koiter E, Racadot S, Abdah-Bortnyak R, Van Limbergen EF, Engelen A, De Brouwer P, Struikmans H, Bartelink H; European Organisation for Research and Treatment of Cancer Radiation Oncology and Breast Cancer Groups. Internal mammary and medial supraclavicular lymph node chain irradiation in stage I-III breast cancer (EORTC 22922/10925): 15-year results of a randomised, phase 3 trial. Lancet Oncol. 2020 Dec;21(12):1602-1610. doi: 10.1016/S1470-2045(20)30472-1. Epub 2020 Nov 2. PMID 33152277
- [Derived] Poortmans PM, Collette S, Kirkove C, Van Limbergen E, Budach V, Struikmans H, Collette L, Fourquet A, Maingon P, Valli M, De Winter K, Marnitz S, Barillot I, Scandolaro L, Vonk E, Rodenhuis C, Marsiglia H, Weidner N, van Tienhoven G, Glanzmann C, Kuten A, Arriagada R, Bartelink H, Van den Bogaert W; EORTC Radiation Oncology and Breast Cancer Groups. Internal Mammary and Medial Supraclavicular Irradiation in Breast Cancer. N Engl J Med. 2015 Jul 23;373(4):317-27. doi: 10.1056/NEJMoa1415369. PMID 26200978